CLINICAL TRIAL: NCT00929279
Title: Facilitation Through Abciximab By drOpping Infusion Line in Patients Undergoing Coronary Stenting. SYNergy With Clopidogrel at High Loading dOse Regimen
Brief Title: Efficacy of Abciximab Bolus Only Regimen in Providing Inhibition of Platelet Action Over Time
Acronym: FABOLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Azienda Ospedaliera Universitaria di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAS-07-I
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2009-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Abciximab; Bolus; Infusion; platelet inhibition; Non ST segment elevation acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abciximab bolus plus infusion (Active Comparator): Abciximab bolus of 0.25mg /Kg, followed by a 12-h infusion 0.125 microg/Kg/min (to a maximum of 10 µg/min) and immediate clopidogrel at 300 mg loading regimen.
  Interventions: Drug: bolus+infusion
- bolus only regimen (Experimental): Abciximab bolus of 0.25mg /Kg followed by placebo infusion and immediate clopidogrel at 600 mg loading dose
  Interventions: Drug: abciximab bolus only regimen

INTERVENTIONS:
Drug: bolus+infusion — Abciximab bolus of 0.25mg /Kg, followed by a 12-h infusion 0.125 microg/Kg/min (to a maximum of 10 µg/min) and immediate clopidogrel at 300 mg loading regimen
  Arms: Abciximab bolus plus infusion
Drug: abciximab bolus only regimen — Abciximab bolus of 0.25mg /Kg followed by placebo infusion and immediate clopidogrel at 600 mg loading dose
  Arms: bolus only regimen

SUMMARY:
In full responders to clopidogrel scheduled to undergo PCI for NSTEACS, the use of abciximab bolus only plus 600 mg clopidogrel loading dose will result in a non-inferior inhibition of platelet aggregation after 4 hours as measured by LTA (20micromol ADP) when compared with abciximab plus infusion and 300 mg clopidogrel loading dose.

DETAILED DESCRIPTION:
Based on the outcome of the EPIC trial, and the sub-optimal results with a single abciximab bolus compared with bolus and infusion, it was recommended to prolong platelet inhibition by a 12h infusion of abciximab after the initial bolus administration in patients undergoing percutaneous coronary intervention (PCI). However, lower outcomes in the single bolus group in the EPIC study were entirely driven by the rates of urgent repeat revascularization at 30 days (3•6 percent bolus group versus 0•8 percent bolus and infusion group, p < 0.001), a complication probably related to the lack of stent use at that time. Importantly, there was no significant difference in terms of death or myocardial infarction (MI). Moreover, the use of clopidogrel in patients undergoing coronary stenting may currently reduce the need for infusion after a single abciximab bolus and it is likely that the soon to come availably of even more potent oral thienopyridines with faster onset of action such as prasugrel may further contribute to make post-bolus abciximab infusion of marginal clinical benefit. Yet, it is known that infusion, as compared to bolus only regimen increases the bleeding rate and the incidence of thrombocytopenia. Thus, bolus only regimen has the potential to maintain protection from ischemic complications in patients undergoing PCI while optimizing the safety profile of the treatment in the current era of intervention based on stents and thienopyridines with fast onset of action.

The CLEAR-PLATELETS study has recently shown that 600 mg clopidogrel does not affect the degree of platelet inhibition throughout infusion of eptifibatide, which is consistent with the notion that glycoprotein IIb/IIIa inhibition at steady state leads to near maximal platelet blockade. No study has so far investigated the effect of clopidogrel, given at high loading dose, in patients treated with abciximab bolus only. In particular, it is not known whether the administration of clopidogrel at high loading dose may prolong the effect of abciximab bolus on the degree of platelet inhibition and if so at which time point the combination of abciximab bolus and clopidogrel may become suboptimal in terms of platelet inhibition as compared to currently recommended 12h infusion of abciximab after the initial bolus administration. This information would lead to relevant clinical implications as it may define the time frame for a safe and effective intervention after bolus only of abciximab in current practice.

This is a single-centre, double-blind prospective randomized pharmacodynamic investigation of 2 antiplatelet regimens in patients undergoing coronary stenting for non-ST segment elevation acute coronary syndromes (NSTECACS):

1. Abciximab bolus followed by infusion plus on-label clopidogrel administration at 300 mg loading dose.
2. abciximab bolus without infusion plus high loading dose of clopidogrel at 600 mg

The objective of the investigation is to test the hypothesis that the administration of abciximab bolus only plus high loading dose of clopidogrel at 600 mg will provide a non inferior level of inhibition of platelet aggregation 4 hours after administration as compared to abciximab bolus followed by standard infusion in combination with clopidogrel loading dose of 300 mg in patients with normal response to clopidogrel (as evaluated after 14-30 days).

ELIGIBILITY:
Inclusion Criteria:

Both of the following:

* Age >18 years
* Symptoms of ischemia that were increasing or occurred at rest, with the last episode occurring no more than 24 hours before randomization;

AND at least one of the following:

* An elevated cardiac troponin T level (≥0.015 μg per liter);
* The presence of ischemic changes as assessed by electrocardiography (defined as ST-segment depression or transient ST-segment elevation exceeding 0.05 mV, or T-wave inversion of ≥0.2 mV in two contiguous leads)
* A documented history of coronary artery disease as evidenced by previous myocardial infarction, findings on previous coronary angiography, or a positive exercise test.

Exclusion Criteria:

* The exclusion criteria are:
* administration of fibrinolytic or any GP IIb IIIa inhibitors for the treatment of current AMI or within 1 month before it
* history of bleeding diathesis
* known sensitivity to abciximab, to any component of the product or to murine monoclonal antibodies
* major surgery or trauma within 30 days
* active bleeding
* previous stroke in the last six months
* oral anticoagulant therapy
* pre-existing thrombocytopenia;
* vasculitis;
* hypertensive retinopathy;
* severe hepatic failure,
* severe renal failure requiring haemodialysis
* documented allergy/intolerance or contraindication to clopidogrel or inability to assume clopidogrel on a consecutive daily basis for a minimum of 30 days, or to heparin or aspirin
* uncontrolled hypertension (systolic or diastolic arterial pressure >180 mmHg or 120, respectively, despite medical therapy)
* limited life expectancy, e.g. neoplasms, others
* inability to obtain informed consent
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
In responders to clopidogrel: Inhibition of platelet aggregation at peak 4h after administration of study drugs measured by LTA (stimulated with 20micromolar ADP) | 4 hours

SECONDARY OUTCOMES:
In all patients treated and in the responders to clopidogrel: • Inhibition of platelet aggregation in the two study groups at time points different from 4 hours after abciximab bolus measured by LTA | up to 24 hours
MACE rate | 30 days
Bleeding rates | 30 days
Thrombocytopenia | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institue of Cardiology, University of Ferrara, Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Valgimigli M, Campo G, Tebaldi M, Monti M, Gambetti S, Scalone A, Parrinello G, Ferrari R; Fabolus Synchro (facilitation through abciximab by dropping infusion Line in patients undergoing coronary stenting. Synergy with clopidogrel at high loading dose regimen) Investigators. Randomized, double-blind comparison of effects of abiciximab bolus only vs. on-label regimen on ex vivo inhibition of platelet aggregation in responders to clopidogrel undergoing coronary stenting. J Thromb Haemost. 2010 Sep;8(9):1903-11. doi: 10.1111/j.1538-7836.2010.03972.x. PMID 20586923